CLINICAL TRIAL: NCT04194892
Title: An Open Label, Randomized, Single Dose, 2-Way Crossover Study to Evaluate the Pharmacokinetics of Pre-filled Syringe Versus Vial Formulations of AM0010 in Healthy Adult Subjects
Brief Title: A Crossover Study to Evaluate Pegilodecakin (LY3500518) in Healthy Participants
Acronym: Willow 3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ARMO BioSciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 17299; J1L-AM-JZGG (Other: Eli Lilly and Company); AM0010-803 (Other: ARMO BioSciences)
Record Dates: First submitted 2019-12-10; First posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Healthy
MeSH Terms: interventions — pegilodecakin; AM0010

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pegilodecakin Vial (Experimental): Pegilodecakin administered subcutaneously (SQ) in one of two study periods.
  Interventions: Biological: Pegilodecakin
- Pegilodecakin Pre-filled syringe (PFS) (Experimental): Pegilodecakin administered SQ in one of two study periods.
  Interventions: Biological: Pegilodecakin

INTERVENTIONS:
Biological: Pegilodecakin — Administered SQ
  Other Names: LY3500518; AM0010

SUMMARY:
The purpose of this study is to assess how fast pegilodecakin gets into the blood stream and how long it takes the body to remove it, when given as a solution formulation via a prefilled syringe (PFS) versus from a vial drawn into a conventional syringe. Information about side effects will be collected. The study is open to healthy participants. Total participant duration in trial is approximately 42 days.

ELIGIBILITY:
Inclusion Criteria:

* Must have a body mass index (BMI) between 19.0 and 32.0 kilograms per meter squared (kg/m²) at study screening
* Must be Human Immunodeficiency Virus (HIV) negative by HIV 1/0/2 testing.
* Must be Hepatitis B (HBV) surface antigen negative
* Must be Hepatitis C (HCV) antibody negative
* Females must have a negative serum pregnancy test

Exclusion Criteria:

* Pregnant or lactating subjects
* Have previously participated in an investigational trial involving administration of any investigational compound within 30 days prior to the study dosing
* Current alcohol or substance abuse judged by the Investigator to potentially interfere with subject compliance
* Have smoked or used tobacco/nicotine products within 90 days prior to the study dosing
* Have been treated with systemic steroids, immunosuppressant therapies or chemotherapeutic agents within 3 months of study screening, or expected to receive these agents during the study (e.g., corticosteroids, immunoglobulins, and other immune- or cytokine-based therapies)
* Have been vaccinated within 90 days of study dosing

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-03-14 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK): Maximum Drug Concentration (Cmax) of Pegilodecakin | Predose through approximately 14 days postdose
  Cmax of Pegilodecakin
PK: Time of Maximum Concentration (Tmax) | Predose through approximately 14 days postdose
  Tmax of Pegilodecakin
PK: Area Under the Serum Concentration Versus Time Curve (AUC) | Predose through approximately 14 days postdose
  AUC of Pegilodecakin

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- PPD Phase 1 Clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No